CLINICAL TRIAL: NCT04609995
Title: Pilot Study of Financial Incentives for YMSM for HIV Testing and PrEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Roland Clayton Merchant, Principal investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020P002907
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: HIV
MeSH Terms: interventions — Fertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No financial incentive (No Intervention): No financial incentives will be provided for completing a PrEP evaluation
- Fixed incentive (Active Comparator): A fixed incentive ($25 Amazon.com gift card) will be provided for completing a PrEP evaluation
  Interventions: Behavioral: Incentives
- Lottery incentive (Active Comparator): An entry into a lottery for a 20% chance to win a $100 Amazon.com gift card will be provided for completing a PrEP evaluation
  Interventions: Behavioral: Incentives

INTERVENTIONS:
Behavioral: Incentives — No financial incentive
  Arms: Fixed incentive; Lottery incentive

SUMMARY:
This pilot, three-arm, randomized trial study involves 200 18-24-year-old young adult men-who-have-sex-with-men (YMSM) recruited through the internet. YMSM are eligible if they are 18-24 years-old, live in the United States, are not known to be HIV infected (self-report), have ever had condomless anal sex with another man, and have never taken HIV pre-exposure prophylaxis (PrEP). The aim of this pilot project is to compare the effect of financial incentives on encouraging YMSM to get tested for HIV and start PrEP for HIV.

Potential study participants will be recruited online through advertising on the internet and complete the study eligibility and consent procedures. Following provision of consent online, participants will be contacted via the email they provided and asked to confirm their willingness to participate. Email addresses are being collected as part of this study to help ensure that individuals do not attempt to participate more than once in this study. Study staff will review the email addresses for duplications. Anyone who attempts to enroll more than once will be disqualified from the study. Participants will not ask for their name as part of the study. Once study interest is confirmed, participants will be provided a study identification number and study arm assignment. They also will be provided with instructions specific to their study arm assignment for the study as well as online resources about HIV testing and PrEP, including options for paying for PrEP.

Participants will be randomly assigned to one of three study arms (no financial incentive, a fixed incentive ($25 Amazon.com gift card) or a lottery (20% for a $100 Amazon.com gift card). Participants in each study arm will be asked to contact the telehealth company PlushCare and make an appointment within two weeks. For this appointment, participants will speak with a PlushCare doctor about being tested for HIV and starting PrEP. They will provide PlushCare with their study identification number. As part of their services, PlushCare will obtain personal identifiers from participants but will not share this information with the study staff.

For this study, participants are asked to undergo an evaluation for PrEP through the PlushCare doctor, but will NOT be required to be tested for HIV nor start PrEP. It will be the participants choice whether or not to be tested for HIV and start or continue PrEP after consultation with the PlushCare doctor. For some participants, the PlushCare doctor might recommend against starting PrEP. PlushCare will follow usual standard-of-care practices for their evaluation, counseling and consideration of PrEP as well as provision and maintenance of services for PrEP. Using only the study identification numbers and not the participant's personal identifiers, PlushCare will provide the study staff with data on completion of the primary and secondary study outcomes.

Participants will be informed that they or their healthcare insurance will bear the costs of HIV testing and PrEP, but not the consultation with PlushCare. They will be provided with resources about how to pay for PrEP from the study as well as PlushCare.

Completion of the primary study outcome (completing an appointment with the telehealth provider PlushCare for a PrEP evaluation) and secondary outcomes (undergoing HIV testing, starting PrEP, time elapsed from study enrollment to PlushCare evaluation, time elapsed to HIV testing and PrEP initiation) will be compared by study arms.

ELIGIBILITY:
Inclusion Criteria: YMSM are eligible if they are 18-24 years-old, live in the United States, are not known to be HIV infected (self-report), have ever had condomless anal sex with another man, and have never taken PrEP.

-

Exclusion Criteria: Not 18-24-years-old, do not live in the US, are known to be HIV infected, have never had condomless anal sex with another man, and have ever taken PrEP

-

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Young adult men-who-have-sex-with-men (YMSM)
Enrollment: 200 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
PrEP evaluation | 30 days
  Completion of PrEP evaluation

IPD SHARING:
Plan to Share IPD: Undecided
Data are intended for a pilot study to support a grant application. Data results and other materials can be obtained upon request after completion of study and analysis.